CLINICAL TRIAL: NCT06890403
Title: Can Stories Encourage the Elderly to Vaccinate? Combining Viewer-tailored Personal Narrative Videos With Informational Videos to Improve Vaccine Uptake Among Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00032331
Record Dates: First submitted 2025-03-20; First posted 2025-03-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Vaccination
Keywords: vaccine; narrative; communication; videos
MeSH Terms: conditions — Narration; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): no videos
- Animation Only (Experimental): informational animation video only
  Interventions: Behavioral: Informational Animation Video
- Narrative Only (Experimental): personal narrative video only
  Interventions: Behavioral: Personal Narrative Video
- Narrative Then Animation (Experimental): personal narrative video followed immediately by the informational animation video
  Interventions: Behavioral: Informational Animation Video; Behavioral: Personal Narrative Video
- Animation Then Narrative (Experimental): informational animation video followed immediately by the personal narrative video
  Interventions: Behavioral: Informational Animation Video; Behavioral: Personal Narrative Video

INTERVENTIONS:
Behavioral: Informational Animation Video — The informational animation video will also take several minutes and will cover human papillomavirus (HPV) disease, address specific concerns when identified, and the importance and safety of HPV vaccines.
  Arms: Animation Only; Animation Then Narrative; Narrative Then Animation
Behavioral: Personal Narrative Video — Personal narrative videos will consist of someone describing the person's own personal experience with HPV. The investigators have a collection of videos of personal narratives from different people that the investigators have cut to approximate several minutes in length so the investigators can tailor the personal narratives to match each study participant's race/ethnicity and gender as closely as possible.
  Arms: Animation Then Narrative; Narrative Only; Narrative Then Animation

SUMMARY:
This study will compare the use of informational videos only, personal story videos only, and the combination of both, to see which is most effective in increasing vaccination among older adults.

ELIGIBILITY:
Inclusion Criteria:

* U.S. adults aged 50 and older

Exclusion Criteria:

* Participants who do not complete the survey
* Participants who are unable or refuse to view and listen to videos on the participant's device

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who receive vaccine | 9-month follow-up
  Vaccination status. Binary variables (received vs not received) for each vaccine recommended for older adults

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Salmon, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Ipsos, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No